CLINICAL TRIAL: NCT04302779
Title: Investigating the Influence of Age and Saliva Flow on the Perception of Protein Fortified Foods and Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Lisa Methven, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 19/67
Record Dates: First submitted 2020-02-11; First posted 2020-03-10 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Individual Difference; Food Sensitivity; Food Preferences
Keywords: Older adults; Oral Nutritional Supplements; Saliva Flow; Mucoadhesion; Mouthdrying
MeSH Terms: conditions — Food Intolerance; Food Preferences

STUDY DESIGN:
Intervention Model Description: This study involves both a crossover design where each participant tastes both the control product (not fortified) and the protein fortified product with an appropriate break between the two sessions. It is also both a within and between groups design as the responses from the older participants will be compared to the younger participants. The study will be conducted single blind as it not feasible to blind the researcher. Each participant will attend 2 study visits and all foods will be presented with random blinding codes.
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solid Model (Experimental): Whey Permeate Lemon Cupcake and Protein Fortified Lemon Cupcake
  Interventions: Behavioral: Solid Model
- Liquid Model (Experimental): Whey Protein Beverage
  Interventions: Behavioral: Liquid Model

INTERVENTIONS:
Behavioral: Solid Model — Cupcakes will be used, with the amount of protein varied to study the effect on perception of the products (using sensory methods rating drying and discrimination tests 'which is the stronger in drying'). Measuring mucoadhesion via protein content remaining in saliva samples following consumption of cupcakes.
  Arms: Solid Model
Behavioral: Liquid Model — To study the perception of whey protein beverages using repeated consumption sensory methods (e.g. rating mouthdrying over repeated sips of the drink).
  Arms: Liquid Model

SUMMARY:
Brief Summary: This study aims to investigate whether protein fortification of foods and beverages causes mouthdrying and mucoadhesion and whether this is influenced by age and saliva flow.

DETAILED DESCRIPTION:
To investigate whether whey protein beverages cause mouthdrying in older adults and if perception and acceptance are influenced by repeated consumption, age and individual differences in saliva flow.

To investigate whether protein fortification of cupcakes causes mouthdrying and if perception and acceptance are influenced by repeated consumption, age and individual differences in saliva flow in a home environment.

To investigate whether mucoadhesion is present within different food models, if sensitivity to mucoadhesion increases with age and to determine if a reduced salivary flow results in strengthened mucoadhesion.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-30 years or over 65 years)
* Healthy

Exclusion Criteria:

* Cognitively impaired
* Allergies, intolerance and special dietary requirements (for example coeliac disease, lactose / gluten intolerance)
* Suffer from diabetes
* Oral surgery
* Stroke
* Smoker
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Mucoadhesion | Change in protein left in mouth over from baseline to after consumption (45s)
  Ex-vivo analysis using cupcakes (whey permeate and whey protein) (expectorated saliva collection to analyse protein for the extent of mucoadhesion)

SECONDARY OUTCOMES:
Mouthdrying from cupcakes | Change in perceived mouthdruing from baseline over consumption (5 minutes)
  Perceived mouth drying from protein fortified lemon cupcake and whey permeate lemon cupcake using data from repeated consumption sensory methods (rating drying on line scales)
Mouthdrying from whey protein beverages | Change in perceived mouthdruing from baseline over consumption (20 minutes)
  Perceived mouth drying from whey protein beverage using data from repeated consumption sensory methods (rating drying on line scales)
Saliva Collection | Days 1 and 2
  Salivary flow rates from unstimulated and stimulated saliva samples
Questionnaire | Day 1
  Dental status, mouth behaviour, attitudes and portion size data via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Bull SP, Hong Y, Khutoryanskiy VV, Parker JK, Faka M, Methven L. Whey protein mouth drying influenced by thermal denaturation. Food Qual Prefer. 2017 Mar;56(Pt B):233-240. doi: 10.1016/j.foodqual.2016.03.008. PMID 28260840
- [Background] Withers CA, Cook MT, Methven L, Gosney MA, Khutoryanskiy VV. Investigation of milk proteins binding to the oral mucosa. Food Funct. 2013 Nov;4(11):1668-74. doi: 10.1039/c3fo60291e. PMID 24092277
- [Background] Affoo RH, Foley N, Garrick R, Siqueira WL, Martin RE. Meta-Analysis of Salivary Flow Rates in Young and Older Adults. J Am Geriatr Soc. 2015 Oct;63(10):2142-51. doi: 10.1111/jgs.13652. Epub 2015 Oct 12. PMID 26456531
- [Background] Gosney M. Are we wasting our money on food supplements in elder care wards? J Adv Nurs. 2003 Aug;43(3):275-80. doi: 10.1046/j.1365-2648.2003.02710.x. PMID 12859786
- [Background] Kennedy O, Law C, Methven L, Mottram D, Gosney M. Investigating age-related changes in taste and affects on sensory perceptions of oral nutritional supplements. Age Ageing. 2010 Nov;39(6):733-8. doi: 10.1093/ageing/afq104. Epub 2010 Sep 22. PMID 20861088
- [Background] Withers CA, Lewis MJ, Gosney MA, Methven L. Potential sources of mouth drying in beverages fortified with dairy proteins: A comparison of casein- and whey-rich ingredients. J Dairy Sci. 2014 Mar;97(3):1233-47. doi: 10.3168/jds.2013-7273. Epub 2014 Jan 17. PMID 24440265